CLINICAL TRIAL: NCT03414008
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 1291583 (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design) in Healthy Male Subjects
Brief Title: This Study Tests How Different Doses of BI 1291583 Are Taken up in the Body and How Well They Are Tolerated
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1397-0001; 2017-002929-38 (EudraCT Number)
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Drug Group (Experimental): Single dose
  Interventions: Drug: BI 1291583
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Matching placebo: Tartaric acid

INTERVENTIONS:
Drug: BI 1291583 — Single dose
  Other Names: Verducatib
  Arms: Active Drug Group
Drug: Matching placebo: Tartaric acid — Single dose
  Arms: Placebo Group

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1291583 in healthy male subjects following oral administration of single rising doses.

Secondary objectives are the exploration of the pharmacokinetics (PK) including dose proportionality and pharmacodynamics (PD) of BI 1291583 after single dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects with WOCBP partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication
* Known relevant immunodeficiency
* Oral body temperature of more than 37.7°C on Day -3 to -1.
* Volunteers who have received live or live-attenuated vaccine in the 4 weeks prior to dosing.
* C-reactive protein above upper limit of laboratory reference range at screening and/or on Day -3 to -1.
* Subjects with signs of current gingivitis/periodontitis. Inspection of the oral cavity will be performed by the investigator
* Subjects with a history of hyperkeratosis or erythema in palms or soles

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability of BI 1291583 is the number [N (%)] of subjects with drug-related adverse events | up to 120 hours

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 120 hours
Cmax (maximum measured concCmax (maximum measured concentration of the analyte in plasma)entration of the analyte in plasma) | up to 120 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com